CLINICAL TRIAL: NCT04297917
Title: A Phase 1 Monotherapy Study to Evaluate the Safety, Tolerability & Immunogenicity of Vaccination With Candidate Chimpanzee Adenovirus-vectored HepB Virus Vaccine ChAdOx1 HBV in Healthy Participants & Participants With Chronic HepB Infection
Brief Title: First in Human Study of ChAdOx1-HBV in Healthy Participants and Participants With Chronic hepB Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBV001
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis B; Healthy
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: The participants were recruited in 6 cohorts as follows - Cohort 1 - Healthy Volunteers - Low dose Vaccine - 5 participants Cohort 2 - Healthy Volunteers - High dose Vaccine - 5 participants Cohort 3 - Participants with Chronic Hepatitis B infection - Low dose - 6 participants Cohort 4 - Participants with Chronic Hepatitis B infection - High dose - 5 participants Cohort 5 - Healthy Volunteers who have completed 2 doses of COVID-19 AZD1222 vaccine Cohort 6 - Healthy Volunteers who have completed 2 doses of either Pfizer or Moderna mRNA COVID 19 vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy Volunteers with low dose vaccination (Experimental): 5 Healthy Volunteers receiving low dose vaccination
  Interventions: Biological: ChAdOx1-HBV
- Healthy Volunteers with high dose vaccination (Experimental): 5 Healthy Volunteers receiving high dose vaccination
  Interventions: Biological: ChAdOx1-HBV
- Chronic Hepatitis B participants with low dose vaccination (Experimental): 6 participants with Chronic Hepatitis B infection receiving low dose vaccination
  Interventions: Biological: ChAdOx1-HBV
- Chronic Hepatitis B participants with high dose vaccination (Experimental): 5 participants with Chronic Hepatitis B infection receiving high dose vaccination
  Interventions: Biological: ChAdOx1-HBV
- Healthy Volunteers who have had COVID-19 AZD1222 vaccine (Experimental): 15 participants who have had 2 doses of COVID-19 AZD1222 vaccine receiving high dose vaccination.
  Interventions: Biological: ChAdOx1-HBV
- Healthy Volunteers who have had Pfizer/Moderna mRNA COVID 19 vaccine (Experimental): 11 participants who have had 2 doses of either Pfizer/Moderna mRNA COVID 19 vaccine receiving high dose vaccination
  Interventions: Biological: ChAdOx1-HBV

INTERVENTIONS:
Biological: ChAdOx1-HBV — chimpanzee adenovirus-vectored hepatitis B virus vaccine

SUMMARY:
This is a Phase 1, first in human study of ChAdOx1-HBV. The study will be conducted in 40 healthy participants and 12 participants with CHB and virally suppressed with oral antiviral medication. This will be an open-label, non randomised dose escalation study comparing the safety, tolerability and immunogenicity of 2 different doses of ChAdOx1 HBV vaccine. T cell responses in healthy participants who have received a prior two-dose series of AZD1222 will be compared with those who have received either the Pfizer COVID 19 vaccine or the Moderna mRNA COVID 19 vaccine.

DETAILED DESCRIPTION:
This is a first in man human study of a therapeutic vaccine for chronic hepatitis B infection(ChAdOx1-1HBV). The vaccine was given to participants in a dose escalation strategy (two doses). Five healthy participants was administered the low dose first (cohort 1). Dose escalation was only initiated in the next 5 healthy participants (cohort 2) following Safety Monitoring Committee (SMC) review.

Six CHB participants was administered the low dose (cohort 3) before the dose escalation was initiated in the remaining 5 CHB participants (cohort 4).

Twenty-six healthy participants (15 who have received two doses of AZD1222 [cohort 5] and 11 who have received at least two prior doses of Pfizer/Moderna mRNA COVID 19 vaccine [cohort 6]) were dosed in parallel with the high dose used in cohorts 2 and 4.

Each participant received 1 dose of the vaccine (intramuscular injection). Participants (Volunteers & patients) in cohorts 1 to 4 attended up to 9 study visits and cohorts 5 & 6 attended up to 4 visits in total. The last visit was 24 weeks after vaccination for cohorts 1 to 4 and 12 weeks for cohorts 5 & 6.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged ≥18 to ≤65 years at screening
2. Body Mass Index ≤30 kg/m2
3. Able to provide informed consent indicating they understand the purpose of, and procedures required, for the study and are willing to participate
4. If female, willing not to become pregnant up to 8 weeks after last dose of study vaccine, not breast feeding
5. If female: Not pregnant, and one of the following:

   * Of non-childbearing potential (i.e. women who have had a hysterectomy or tubal ligation or are post menopausal, as defined by no menses in ≥1 year)
   * Sexual abstinence, only if the participant refrains from heterosexual intercourse during the entire study period and it is the usual lifestyle of the participant
   * Of childbearing potential but agrees to practice highly effective contraception for 4 weeks prior to study vaccine and 8 weeks after study vaccine. Highly effective methods of contraception include one or more of the following:

   Male partner who is sterile (medically effective vasectomy) prior to the female participant's entry into the study and is the sole sexual partner for the female participant, Hormonal (oral, intravaginal, transdermal, implantable or injectable), An intrauterine hormone releasing system, An intrauterine device and Bilateral tubal occlusion

   Healthy participants (cohorts 1 and 2):
6. Considered to be healthy with no current conditions that may significantly impair participant safety or influence study results, in the opinion of the Investigator

   Participants with well controlled CHB (cohorts 3 and 4):
7. Documented evidence of chronic HBV infection (e.g. HBsAg positive ≥6 months with detectable HBsAg levels at screening)
8. Receipt of only either entecavir or tenofovir for at least 12 months before screening
9. Virally suppressed (HBV DNA <40 IU/mL for ≥6 months)
10. HBsAg <4000IU/mL

Participants with well controlled CHB (cohorts 3 and 4):

7. Documented evidence of chronic HBV infection (e.g. HBsAg positive ≥6 months with detectable HBsAg levels at screening) 8. Receipt of only either entecavir or tenofovir for at least 12 months before screening 9. Virally suppressed (HBV DNA <40 IU/mL for ≥6 months) 10. HBsAg <10000 IU/mL

Healthy participants (cohort 5):

11. Considered to be healthy with no current conditions that may significantly impair participant safety or influence study results, in the opinion of the Investigator 12. Adult males or females aged ≥40 to ≤60 years at screening 13. Completed second dose of COVID-19 AZD1222 vaccine 10 to 18 weeks before enrolment

Healthy participants (cohort 6):

14. Considered to be healthy with no current conditions that may significantly impair participant safety or influence study results, in the opinion of the Investigator

15. Adult males or females aged ≥40 to ≤60 years at screening

16. Received the latest dose of Completed of either Pfizer (Comirnaty®) or Moderna (Spikevax) mRNA COVID 19 vaccine 6 to 30 weeks before enrolment

Exclusion Criteria:

1. Presence of any significant acute or chronic, uncontrolled medical/ psychiatric illness
2. Hepatitis C virus antibody positive.
3. Human immunodeficiency virus antibody positive
4. History or evidence of autoimmune disease or known immunodeficiency of any cause
5. Prolonged therapy with immunomodulators (e.g. corticosteroids) or biologics (e.g. monoclonal antibodies, interferon) within 3 months of screening
6. Receipt of immunoglobulin or other blood products within 3 months prior to screening
7. Receipt of any investigational drug or vaccine within 3 months prior to screening
8. Cohorts 1-4: Receipt of any adenoviral vaccine within 3 months prior to administration of ChAdOx1-HBV on Day 0, or plan to receive an adenoviral-based vaccine within 3 months after Day 0

   Cohorts 5 and 6: Receipt of any adenoviral vaccine (other than AZD1222 per inclusion criterion 13) within 3 months prior to administration of ChAdOx1-HBV on Day 0, or plan to receive an adenoviral-based vaccine within 3 months after Day 0
9. Receipt of any live vaccines within 30 days prior to screening
10. Receipt of any inactivated vaccines within 14 days prior to screening
11. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
12. Any history of anaphylaxis in reaction to vaccination
13. Malignancy within 5 years prior to screening with the exception of specific cancers that are cured by surgical resection (e.g. except basal cell skin carcinoma of the skin and cervical carcinoma). Participants under evaluation for possible malignancy are not eligible
14. Current alcohol or substance abuse judged by the Investigator to potentially interfere with participant safety and compliance
15. Significant cardiac disease or unstable uncontrolled cardiac disease
16. Any laboratory test at screening which is abnormal and which is deemed by the Investigator to be clinically significant
17. Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study Additionally, for healthy participants (cohorts 1, 2, 5 and 6)
18. HBsAg positive Additionally, for participants with well controlled CHB (cohorts 3 and 4)
19. Co infection with hepatitis delta
20. Documented cirrhosis or advanced fibrosis indicated by a liver biopsy within 6 months prior to screening.

    In the absence of an appropriate liver biopsy, either 1 of the following:
    * Screening Fibroscan with a result >9 kPa within ≤6 months of screening or
    * Screening FibroTest >0.48 and aspartate aminotransferase (AST) to platelet ratio index of >1 In the event of discordant results between non-invasive methods, the Fibroscan result will take precedence.
21. Alanine transaminase (ALT) >3 × upper limit of normal, international normalised ratio (INR) >1.5 unless the participant was stable on an anticoagulant regimen affecting INR, albumin <35 g/L, total bilirubin >2 mg/dL, platelet count <100,000/mL
22. A history of liver decompensation (e.g. ascites, encephalopathy or variceal haemorrhage)
23. Prior or current hepatocellular carcinoma
24. Chronic liver disease of a non HBV aetiology
25. Any herbal supplements and or other medicines with potential liver toxicity within the previous 3 months prior to enrolment into this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Barnes, Prof, Principal Investigator — University of Oxford
Locations (4):
- United Kingdom (4):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Oxford University Hospitals Nhs Foundation Trust, Oxford, Oxfordshire
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Headington, Oxford
  - Medicines Evaluations Unit, Manchester

REFERENCES:
- [Derived] Cargill T, Cicconi P, Brown A, Holland L, Karanth B, Rutkowski K, Ashwin E, Mehta R, Chinnakannan S, Sebastian S, Bussey L, Sorensen H, Klenerman P, Evans T, Barnes E. HBV001: Phase I study evaluating the safety and immunogenicity of the therapeutic vaccine ChAdOx1-HBV. JHEP Rep. 2023 Aug 18;5(11):100885. doi: 10.1016/j.jhepr.2023.100885. eCollection 2023 Nov. PMID 37791379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-seven (57) participants were screened. Forty-seven (47) subjects were enrolled and vaccinated. The study consisted of 36 healthy participants and 11 participants with CHB and virally suppressed with oral antiviral medication.
Groups:
- Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination: 15 participants who have had 2 doses of COVID-19 AZD1222 vaccine
  ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination: 11 participants who have had Pfizer/Moderna mRNA COVID 19 vaccine
  ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
Period: Overall Study
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Started | 5 | 5 | 6 | 5 | 15 | 11
Completed | 5 | 4 | 6 | 5 | 15 | 11
Not Completed | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine: 15 participants who have had 2 doses of COVID-19 AZD1222 vaccine
  ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine: 11 participants who have had Pfizer/Moderna mRNA COVID 19 vaccine
  ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine | Total
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 15 | 11 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (7.92) | 38.0 (5.15) | 39.0 (7.51) | 40.8 (5.63) | 50.1 (6.62) | 50.3 (6.92) | 45.2 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 7 | 6 | 21
  Male | 4 | 3 | 4 | 2 | 8 | 5 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 3 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 1 | 1 | 4
  White | 4 | 5 | 3 | 0 | 12 | 10 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Height at Screening [Mean (Standard Deviation); unit: cm] | 173.70 (1.107) | 172.92 (5.814) | 175.00 (11.967) | 162.20 (15.515) | 172.34 (11.864) | 170.94 (8.344) | 171.48 (10.467)
Weight at Screening [Mean (Standard Deviation); unit: kg] | 71.18 (9.030) | 76.80 (7.661) | 69.50 (10.766) | 63.26 (16.646) | 76.65 (12.988) | 74.91 (8.975) | 73.34 (11.691)
BMI at Screening [Mean (Standard Deviation); unit: kg/m^2] | 23.60 (2.983) | 25.62 (1.377) | 22.65 (2.669) | 23.74 (3.135) | 25.77 (2.866) | 25.66 (2.862) | 24.88 (2.877)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Safety and Reactogenicity Events: Adverse Events
Description: Adverse events and/or adverse events leading to study discontinuation. Percentages are based on the number of participants in the Safety Analysis Set.
Time Frame: Recorded in the eCRF from the date the informed consent is signed, at all clinic visits (D0, D1, D7, D14, D28, D56, D84) to cover the period since the previous visit and during the visit and up to 168 days post-vaccination (6 months)
Population: Safety analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 15 | 11
Participants
  Number of Participants with any Adverse Event | 1 | 4 | 2 | 4 | 8 | 8
  Number of Participants with Adverse Event leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Incidence of Safety and Reactogenicity Events: Serious Adverse Events
Description: Serious adverse events related to the study vaccine. Percentages are based on the number of participants in the Safety Analysis Set.
Time Frame: From day 0 to up to 6 months
Population: Safety Analysis Set - all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 15 | 11
Participants
  Participants experiencing Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0
  No Events | 5 | 5 | 6 | 5 | 15 | 11

3. Primary Outcome: Incidence of Safety and Reactogenicity Events: Grade ≥3 Local Reactions
Description: Local reactions were collected by the investigator pre and post vaccination on Day 0. In addition, local reactions were captured in the participant diary card on Days 1, 2 and 3. The number and percentage of participants who experienced any symptom are summarised.
Time Frame: From day 0 to day 3
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 15 | 11
participants
  Swelling - Grade ≥3 Local reactions | 0 | 0 | 0 | 0 | 0 | 0
  Redness - Grade ≥3 Local reactions | 0 | 0 | 0 | 0 | 0 | 0
  Pain - Grade ≥3 Local reactions | 0 | 0 | 0 | 0 | 0 | 0
  Warmth - Grade ≥3 Local reactions | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Safety and Reactogenicity Events: Grade ≥3 Systemic Reactions
Description: Systemic reactions were collected by the investigator pre and post vaccination on Day 0 and captured in the participant diary card on Days 1, 2 and 3. The number and percentage of participants who experienced any symptom are summarised.
Time Frame: From day 0 to day 3
Population: Safety Analysis Sets
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 15 | 11
Participants
  Temperature: 0 = None | 5 | 4 | 6 | 5 | 15 | 11
  Temperature: 1 = No interference with daily activities | 0 | 1 | 0 | 0 | 0 | 0
  Temperature: 2 = Some interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Ache: 0 = None | 4 | 1 | 3 | 3 | 12 | 3
  Muscle Ache: 1 = No interference with daily activities | 1 | 1 | 2 | 0 | 3 | 6
  Muscle Ache: 2 = Some interference with daily activities | 0 | 3 | 1 | 2 | 0 | 2
  Muscle Ache: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Ache: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue: 0 = None | 4 | 4 | 3 | 3 | 14 | 6
  Fatigue: 1 = No interference with daily activities | 0 | 1 | 2 | 0 | 1 | 3
  Fatigue: 2 = Some interference with daily activities | 1 | 0 | 1 | 2 | 0 | 2
  Fatigue: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Headache: 0 = None | 5 | 4 | 5 | 4 | 15 | 8
  Headache: 1 = No interference with daily activities | 0 | 0 | 0 | 0 | 0 | 1
  Headache: 2 = Some interference with daily activities | 0 | 1 | 1 | 1 | 0 | 2
  Headache: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Headache: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: 0 = None | 5 | 5 | 5 | 4 | 15 | 11
  Nausea: 1 = No interference with daily activities | 0 | 0 | 1 | 0 | 0 | 0
  Nausea: 2 = Some interference with daily activities | 0 | 0 | 0 | 1 | 0 | 0
  Nausea: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Feverishness: 0 = None | 5 | 4 | 4 | 5 | 15 | 11
  Feverishness: 1 = No interference with daily activities | 0 | 0 | 1 | 0 | 0 | 0
  Feverishness: 2 = Some interference with daily activities | 0 | 1 | 1 | 0 | 0 | 0
  Feverishness: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Feverishness: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Chills: 0 = None | 5 | 4 | 6 | 4 | 14 | 10
  Chills: 1 = No interference with daily activities | 0 | 0 | 0 | 1 | 1 | 0
  Chills: 2 = Some interference with daily activities | 0 | 1 | 0 | 0 | 0 | 1
  Chills: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Chills: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Joint Ache: 0 = None | 5 | 4 | 5 | 4 | 14 | 10
  Joint Ache: 1 = No interference with daily activities | 0 | 0 | 1 | 1 | 1 | 0
  Joint Ache: 2 = Some interference with daily activities | 0 | 1 | 0 | 0 | 0 | 1
  Joint Ache: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Joint Ache: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: 0 = None | 5 | 4 | 5 | 4 | 15 | 9
  Malaise: 1 = No interference with daily activities | 0 | 1 | 0 | 0 | 0 | 2
  Malaise: 2 = Some interference with daily activities | 0 | 0 | 1 | 1 | 0 | 0
  Malaise: 3 = Significant interference with daily activities | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: 4 = ER visit or hospitalisation | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Effect of Prior AZD1222 on the CD8+ T Cell Magnitude and Phenotype as Measured by Multiparameter Flow Cytometry
Description: Intracellular cytokine staining analysis to measure IFNγ, produced by HBV antigen or hexon-specific CD8+ T cells in PBMC across study timepoints
Time Frame: Baseline, Day 14, 28, 56, 84
Reporting Status: Not Posted

6. Secondary Outcome: Reduction in HBsAg Titre Post-vaccination in CHB Participants
Description: For the CHB participants only. HBsAg levels were measured at each scheduled follow-up timepoint (Day 28, Day 56, Day 84 and Day 168).
  A summary of the change is obtained by summarising the difference in the log-transformed results [log(HbsAg at baseline + 1) - log(HbsAg at follow-up + 1)] and back-transforming to absolute values (IU/mL). The mean change is then the Geometric Mean (GM) ratio, where a GM ratio > 1 is equivalent to a reduction in HbsAg.
Time Frame: Baseline, Day 28, 56, 84 and 168
Population: Per Protocol population used for HBsAg changes
Measure: Geometric Mean (Standard Deviation); unit: ratio
Groups:
- Chronic Hepatitis B Participants With Low Dose Vaccination: 6 participants with Chronic Hepatitis B infection receiving low dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Chronic Hepatitis B Participants With High Dose Vaccination: 5 participants with Chronic Hepatitis B infection receiving high dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
Arm/Group | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination
Number analyzed (Participants) | 6 | 5
ratio
  Day 28 | 1.019 (1.1569) | 0.957 (1.0760)
  Day 56 | 1.086 (1.3271) | 0.814 (1.4126)
  Day 84 | 0.984 (1.3271) | 0.901 (1.1471)
  Day 168 | 1.418 (1.5074) | 1.055 (1.0857)

7. Secondary Outcome: Loss of Both HBeAg and HBsAg
Description: For the CHB participants only, loss of HBeAg and HBsAg at the End of Study assessment (Day 168) include all CHB participants in the denominator. Numerators include participants with a) detectable HBeAg and HBsAg at the Day 0 pre-dose assessment and b) undetectable HBeAg and HBsAg at the End of Study assessment.
Time Frame: Baseline and Day 168
Population: Intent to Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination
Number analyzed (Participants) | 6 | 5
Participants
  Yes (loss of both HBeAg and HBsAg) | 0 | 0
  No | 6 | 5

8. Secondary Outcome: Proportion of CHB Participants With HBeAg and HBsAg Seroconversion
Description: The seroconversion of HBeAg and HBsAg is defined as loss of response to the antigen (defined as a value below the limit of detection (i.e. Not detected) and development of antibody to either HBeAg or surface antigen (HBsAg) (defined as a measurable value above the limit of detection (i.e. Detected). The number and percentage of CHB participants meeting the criteria for seroconversion will be summarised.
Time Frame: Baseline, Day 28, 56, 84 and 168
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination
Number analyzed (Participants) | 6 | 5
Participants
  HBsAg Seroconversion: Seroconversion | 0 | 0
  HBsAg Seroconversion: No Seroconversion | 6 | 5
  HBeAg Seroconversion: Seroconversion | 0 | 0
  HBeAg Seroconversion: No Seroconversion | 6 | 5

9. Secondary Outcome: Reduction of Hepatitis B DNA Levels in CHB Participants
Description: Change in hepatitis B DNA levels is defined by subtracting the DNA levels at each follow-up visit (Day 28, Day 56, Day 84 and Day 168) from the DNA levels pre-vaccination (Day 0). A positive change is equivalent to a reduction in DNA levels. Any results recorded as Not Detected were replaced with zero prior to summarising while any recorded as Detected or 1 (the limit of detection) were replaced with 0.5, prior to summarising. The denominator is the number of participants in the analysis set.
Time Frame: Baseline, Day 28, 56, 84 and 168
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: log 10 IU/ml
Arm/Group | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination
Number analyzed (Participants) | 6 | 5
log 10 IU/ml
  Baseline | 0.000 (0.000) | 0.432 (0.5942)
  Day 28 | -0.333 (0.4082) | 0.156 (1.0159)
  Day 56 | -0.455 (0.5500) | 0.432 (0.5942)
  Day 84 | -0.425 (0.5037) | 0.198 (0.9379)
  Day 168 | -0.333 (0.5164) | 0.032 (0.7649)

10. Secondary Outcome: Percentage of CD4+ and CD8+ Expressing IFNγ at Baseline and Days 14, 28, 56, and 84 After Vaccination
Description: CD4+ and CD8+ cells were analyzed at selected baseline and follow up study visits (Day 0, Day 14, Day 28, Day 56, and/or Day 84) using intracellular cytokine staining (ICS) data from a flow cytometer. Outcome 'A Multiparameter Index Made of CD4+Magnitude, CD4+ Avidity and CD8+ Magnitude' was not calculated.
Time Frame: Baseline, 14, 28, 56, and 84
Population: The intention was to correlate the measure to hep B surface antigen response, which was not observed any group. We report available data for CD4+ and CD8+ magnitude from Groups 1, 2, 5, and 6. ICS assays were performed at baseline and at the timepoint of peak total response magnitude where adequate cell numbers were available (Baseline and Day 14, 28, 56, and/or 84 after dosing). No results obtained for Groups 3 and 4 due to insufficient sample volume. Certain time points were not collected.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Groups:
- Group 1 Healthy Volunteers With Low Dose Vaccination: 5 Healthy Volunteers receiving low dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Group 2 Healthy Volunteers With High Dose Vaccination: 5 Healthy Volunteers receiving high dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Group 3 Chronic Hepatitis B Participants With Low Dose Vaccination: 6 participants with Chronic Hepatitis B infection receiving low dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Group 4 Chronic Hepatitis B Participants With High Dose Vaccination: 5 participants with Chronic Hepatitis B infection receiving high dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Group 5 Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination: 15 participants who have had 2 doses of COVID-19 AZD1222 vaccine ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Group 6 Healthy Volunteers Who Have Had mRNA COVID 19 Vaccine Received High Dose Vaccination: 11 participants who have had Pfizer/Moderna mRNA COVID 19 vaccine ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
Arm/Group | Group 1 Healthy Volunteers With Low Dose Vaccination | Group 2 Healthy Volunteers With High Dose Vaccination | Group 3 Chronic Hepatitis B Participants With Low Dose Vaccination | Group 4 Chronic Hepatitis B Participants With High Dose Vaccination | Group 5 Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Group 6 Healthy Volunteers Who Have Had mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 0 | 0 | 15 | 10
Percentage of cells
  CD4+ (Day 0): number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 9
  CD4+ (Day 0) |  |  |  |  | 0.019 (0.021) | 0.016 (0.013)
  CD4+ (Day 14) | 0.013 (0.013) | 0.013 (0.013) |  |  | 0.015 (0.016) | 0.048 (0.037)
  CD4+ (Day 28) | 0.013 (0.003) | 0.005 (0.000) |  |  | 0.017 (0.013) | 0.054 (0.042)
  CD4+ (Day 56): number analyzed (Participants) | 5 | 5 | 0 | 0 | 0 | 0
  CD4+ (Day 56) | 0.001 (0.000) | 0.023 (0.011) |  |  |  |
  CD4+ (Day 84): number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 9
  CD4+ (Day 84) |  |  |  |  | 0.020 (0.015) | 0.033 (0.025)
  CD8+ (Day 0): number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 9
  CD8+ (Day 0) |  |  |  |  | 0.055 (0.085) | 0.076 (0.109)
  CD8+ (Day 14) | 0.022 (0.014) | 0.072 (0.044) |  |  | 0.073 (0.125) | 1.319 (3.685)
  CD8+ (Day 28) | 0.046 (0.022) | 0.000 (0.000) |  |  | 0.063 (0.074) | 2.365 (7.406)
  CD8+ (Day 56): number analyzed (Participants) | 5 | 5 | 0 | 0 | 0 | 0
  CD8+ (Day 56) | 0.293 (0.000) | 0.089 (0.073) |  |  |  |
  CD8+ (Day 84): number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 9
  CD8+ (Day 84) |  |  |  |  | 0.058 (0.059) | 7.148 (23.172)

11. Secondary Outcome: Total T Cell Response to the Core Antigen Encoded by ChAdOx1-HBV as Measured in a Peptide-stimulated ELISpot Assay
Description: This was determined by using PMBCs in IFN-γ ELISpot assays to investigate the breadth of HBV specific T cell responses. Assessment of immune response was based on the number of IFN-γ spot-forming units (SFU) per 10^6 PBMC in response to stimulation with each antigenic peptide pool. For CHB-LD, CHB-HD, HP-LD, HP-HD the background correction is derived by subtracting the relevant DMSO control result and replacing any negative values or values < 25 with zero prior to summarising.
Time Frame: Baseline, Day 14, 28, 56, 84 and 168
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: Spot forming units (SFU) per 10^6 PBMC
Groups:
- Healthy Volunteers With Low Dose Vaccination: 5 Healthy Volunteers receiving low dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
- Healthy Volunteers With High Dose Vaccination: 5 Healthy Volunteers receiving high dose vaccination ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 14 | 11
Spot forming units (SFU) per 10^6 PBMC
  Baseline: number analyzed (Participants) | 5 | 2 | 5 | 5 | 14 | 11
  Baseline | 30.00 (67.0820) | 0.000 (0.000) | 0.000 (0.0000) | 18.200 (27.2250) | 16.111 (32.4286) | 40.000 (70.0317)
  Day 14: number analyzed (Participants) | 5 | 1 | 5 | 5 | 14 | 11
  Day 14 | 148.067 (33.5090) | 135.000 (0.000) | 17.000 (26.3629) | 33.800 (52.9925) | 62.341 (72.5715) | 162.727 (222.4751)
  Day28: number analyzed (Participants) | 5 | 1 | 5 | 5 | 14 | 11
  Day28 | 225.667 (161.5661) | 181.667 (0.000) | 39.600 (88.5483) | 31.400 (70.2125) | 51.507 (107.5817) | 96.969 (109.7602)
  Day 56: number analyzed (Participants) | 5 | 1 | 5 | 5 | 0 | 0
  Day 56 | 99.833 (66.5061) | 76.667 (0.000) | 5.000 (11.1803) | 81.600 (83.7425) |  |
  Day 84: number analyzed (Participants) | 5 | 1 | 5 | 5 | 13 | 11
  Day 84 | 66.333 (81.8739) | 0.000 (0.000) | 0.000 (0.0000) | 43.060 (71.5616) | 113.075 (205.7545) | 60.302 (65.6994)
  Day 168: number analyzed (Participants) | 5 | 1 | 5 | 5 | 0 | 0
  Day 168 | 49.667 (68.3171) | 38.333 (0.000) | 6.000 (13.4164) | 14.200 (31.7522) |  |

12. Secondary Outcome: Total T Cell Response to the Pol1-Pol4 Antigen Encoded by ChAdOx1-HBV as Measured in a Peptide-stimulated ELISpot Assay
Description: as for outcome 11
Time Frame: Baseline, Day 14, 28, 56, 84 and 168
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: Spot forming units (SFU) per 10^6 PBMC
Groups:
- Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination: 14 participants who have had 2 doses of COVID-19 AZD1222 vaccine ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 15 | 11
Spot forming units (SFU) per 10^6 PBMC
  Baseline: number analyzed (Participants) | 5 | 2 | 5 | 5 | 14 | 11
  Baseline | 61.000 (87.4929) | 22.500 (31.8198) | 6.200 (13.8636) | 11.600 (25.9384) | 0.000 (0.000) | 0.000 (0.000)
  Day 14: number analyzed (Participants) | 5 | 1 | 5 | 5 | 14 | 11
  Day 14 | 459.600 (190.4637) | 680.000 (0.000) | 64.000 (95.8775) | 13.000 (29.0689) | 15.317 (39.9482) | 252.727 (347.2137)
  Day 28: number analyzed (Participants) | 5 | 1 | 5 | 5 | 14 | 11
  Day 28 | 585.333 (207.7338) | 853.333 (0.000) | 102.200 (206.8918) | 44.600 (85.9349) | 5.238 (19.5992) | 134.090 (203.8124)
  Day 56: number analyzed (Participants) | 5 | 1 | 5 | 5 | 0 | 0
  Day 56 | 143.333 (94.4410) | 670.000 (0.000) | 55.800 (103.8663) | 130.000 (262.5871) |  |
  Day 84: number analyzed (Participants) | 5 | 1 | 5 | 5 | 13 | 11
  Day 84 | 254.000 (142.9773) | 385.000 (0.000) | 74.000 (111.2654) | 15.600 (34.8827) | 40.513 (122.9345) | 68.485 (124.9477)
  Day 168: number analyzed (Participants) | 5 | 1 | 5 | 5 | 0 | 0
  Day 168 | 209.333 (144.9119) | 260.833 (0.000) | 0.000 (0.0000) | 7.000 (15.6525) |  |

13. Secondary Outcome: Total T Cell Response to the Pre S1/S2 Surface Antigen Encoded by ChAdOx1-HBV as Measured in a Peptide-stimulated ELISpot Assay
Description: as for outcome 11
Time Frame: Baseline, Day 14, 28, 56, 84 and 168
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: Spot forming units (SFU) per 10^6 PBMC
Groups:
- Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Vaccination: 11 participants who have had Pfizer/Moderna mRNA COVID 19 vaccine ChAdOx1-HBV: chimpanzee adenovirus-vectored hepatitis B virus vaccine
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 14 | 11
Spot forming units (SFU) per 10^6 PBMC
  Baseline: number analyzed (Participants) | 5 | 3 | 5 | 5 | 14 | 11
  Baseline | 279.167 (296.0316) | 10.000 (17.3205) | 38.200 (70.8110) | 20.200 (31.2282) | 46.349 (76.7025) | 86.364 (101.3734)
  Day 14: number analyzed (Participants) | 5 | 2 | 5 | 5 | 14 | 11
  Day 14 | 613.967 (195.7494) | 918.750 (429.5674) | 32.000 (19.0263) | 35.400 (50.2076) | 94.444 (100.6059) | 191.818 (124.9388)
  Day 28: number analyzed (Participants) | 5 | 2 | 5 | 5 | 14 | 11
  Day 28 | 691.167 (164.1345) | 723.750 (121.9759) | 25.600 (57.2433) | 5.000 (11.1803) | 77.698 (88.9171) | 163.787 (108.5050)
  Day 56: number analyzed (Participants) | 5 | 2 | 5 | 5 | 0 | 0
  Day 56 | 385.000 (173.8813) | 873.333 (546.8292) | 25.400 (26.1878) | 109.600 (220.7788) |  |
  Day 84: number analyzed (Participants) | 5 | 2 | 5 | 5 | 13 | 11
  Day 84 | 341.333 (147.7958) | 348.750 (113.7263) | 32.600 (51.2133) | 19.660 (27.2365) | 100.256 (174.3531) | 79.394 (76.1256)
  Day 168: number analyzed (Participants) | 5 | 2 | 5 | 5 | 0 | 0
  Day 168 | 229.000 (142.8947) | 353.333 (124.9222) | 24.800 (36.7859) | 12.200 (17.1523) |  |

14. Secondary Outcome: Total T Cell Response to the Sii Surface Antigen Encoded by ChAdOx1-HBV as Measured in a Peptide-stimulated ELISpot Assay
Description: as for outcome 11
Time Frame: Baseline, Day 14, 28, 56, 84 and 168
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: Spot forming units (SFU) per 10^6 PBMC
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Vaccination
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 14 | 11
Spot forming units (SFU) per 10^6 PBMC
  Baseline: number analyzed (Participants) | 4 | 0 | 6 | 5 | 0 | 0
  Baseline | 12.500 (25.0000) |  | 0.000 (0.0000) | 5.600 (12.5220) |  |
  Day 14: number analyzed (Participants) | 4 | 0 | 6 | 5 | 0 | 0
  Day 14 | 179.042 (285.1818) |  | 5.600 (12.5220) | 0.000 (0.0000) |  |
  Day 28: number analyzed (Participants) | 4 | 0 | 6 | 5 | 0 | 0
  Day 28 | 322.500 (506.5872) |  | 0.000 (0.0000) | 5.000 (11.1803) |  |
  Day 56: number analyzed (Participants) | 4 | 0 | 6 | 5 | 0 | 0
  Day 56 | 98.750 (197.5000) |  | 0.000 (0.0000) | 38.000 (84.9706) |  |
  Day 84: number analyzed (Participants) | 4 | 0 | 6 | 5 | 0 | 0
  Day 84 | 119.583 (239.1667) |  | 0.000 (0.0000) | 0.000 (0.0000) |  |
  Day 168: number analyzed (Participants) | 4 | 0 | 6 | 5 | 0 | 0
  Day 168 | 91.250 (182.5000) |  | 0.000 (0.0000) | 0.000 (0.0000) |  |

15. Secondary Outcome: Effect of Prior AZD1222 on the CD4+ T Cell Magnitude and Phenotype as Measured by Multiparameter Flow Cytometry
Description: Intracellular cytokine staining analysis to measure IFNγ, produced by hexon-specific CD4+ T cells in PBMC across study timepoints
Time Frame: Baseline, Day 14, 28, 84
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: Mean CD4+ IFNy+ T cells
Arm/Group | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 15 | 11
Mean CD4+ IFNy+ T cells
  CD4+ IFNy+ Day 0 | 0.018525 (0.02152) | 0.016409 (0.014048)
  CD4+ IFNy+ Day 14 | 0.014959 (0.016946) | 0.047705 (0.03924)
  CD4+ IFNy+ Day 28 | 0.017065 (0.013149) | 0.054382 (0.04386)
  CD4+ IFNy+ Day 84 | 0.020178 (0.015547) | 0.033339 (0.026769)

16. Secondary Outcome: Effect of Prior AZD1222 on the CD8+ T Cell Magnitude and Phenotype as Measured by Multiparameter Flow Cytometry
Description: Intracellular cytokine staining analysis to measure IFNγ, produced by hexon-specific CD8+ T cells in PBMC across study timepoints
Time Frame: Baseline, Day 14, 28, 84
Population: Immunogenicity Analysis Set
Measure: Mean (Standard Deviation); unit: Mean CD8+ IFNy+ T cells
Arm/Group | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
Number analyzed (Participants) | 15 | 1
Mean CD8+ IFNy+ T cells
  CD8+ IFNy+ Day 0 | 0.055028 (0.088611) | 0.085174 (0.130337)
  CD8+ IFNy+ Day 14 | 0.073259 (0.129767) | 0.295344 (0.506428)
  CD8+ IFNy+ Day 28 | 0.062521 (0.076278) | 0.261003 (0.34742)
  CD8+ IFNy+ Day 84 | 0.057933 (0.061425) | 0.183798 (0.145222)

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events will be recorded in the eCRF from the date the informed consent is signed, at all clinic visits (D0, D1, D7, D14, D28, D56, D84) to cover the period since the previous visit and during the visit and up to 168 days post-vaccination (6 months). Unsolicited adverse events will be followed until resolved or until participant contact discontinues.
Description: Adverse events were coded using MedDRA. Treatment-emergent adverse events (TEAEs) are defined as those occurring or worsening after the study vaccine administration. TEAEs are summarised by system organ class (SOC) and by preferred term (PT). The incidence of TEAEs is based on the numbers and percentages of participants with events and number of events. TEAEs are further summarised by severity and relationship to study vaccine.
Arm/Group | Healthy Volunteers With Low Dose Vaccination | Healthy Volunteers With High Dose Vaccination | Chronic Hepatitis B Participants With Low Dose Vaccination | Chronic Hepatitis B Participants With High Dose Vaccination | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/5 | 0/15 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/5 | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 1/5 | 4/5 | 2/6 | 4/5 | 8/15 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers With Low Dose Vaccination (N=5) | Healthy Volunteers With High Dose Vaccination (N=5) | Chronic Hepatitis B Participants With Low Dose Vaccination (N=6) | Chronic Hepatitis B Participants With High Dose Vaccination (N=5) | Healthy Volunteers Who Have Had COVID-19 AZD1222 Vaccine Received High Dose Vaccination (N=15) | Healthy Volunteers Who Have Had Pfizer/Moderna mRNA COVID 19 Vaccine Received High Dose Vaccination (N=11)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythrma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laparoscopic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
[Not specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04297917/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04297917/SAP_001.pdf